CLINICAL TRIAL: NCT06626412
Title: Longitudinal Imaging of Striatal Synaptic Density and Volume in People With Premanifest Huntington's Disease.
Brief Title: Longitudinal SV2A and MRI in Premanifest HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S69109
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease
Keywords: PET; MRI; SV2A; synaptic density; 18F-SynVesT-1
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premanifest HD (Experimental): At baseline and 2-year follow-up
  Interventions: Diagnostic Test: Diagnostic Test: 18F-SynVesT-1 PET; Diagnostic Test: Volumetric MRI
- Healthy controls (Active Comparator): At baseline and 2-year follow-up
  Interventions: Diagnostic Test: Diagnostic Test: 18F-SynVesT-1 PET; Diagnostic Test: Volumetric MRI

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: 18F-SynVesT-1 PET — Positron Emission Tomography (PET) of synaptic vesicle protein 2A (SV2A) using the radioligand 18F-SynVesT-1.
Diagnostic Test: Volumetric MRI — Magnetic resonance imaging of brain volume.

SUMMARY:
AIM: to compare the sensitivity of SV2A PET and volumetric MRI to detect longitudinal striatal changes in premanifest HD.

DESIGN: The investigators will include late premanifest HD mutations carriers and matched healthy controls. All subjects will undergo a clinical examination, with comprehensive assessment of motor and non-motor symptoms, and imaging evaluation consisting of 18F-SynVesT-1 PET and volumetric MRI at baseline and after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years inclusive.
* Capacity to understand the informed consent form.
* HD mutation carriers:

  * HTT (CAG)n ≥ 40
  * HD-ISS < 2
  * CAP100 score > 70

Exclusion Criteria:

* neuropsychiatric diseases (other than HD for HD mutation carriers)
* major internal medical diseases
* white matter lesion load on FLAIR Fazekas score 2 or higher or other relevant MRI abnormalities
* history of alcohol abuse or current alcohol abuse (chronic use of more than 15 units per week) or drug abuse
* contraindications for MR
* pregnancy
* previous participation in other research studies involving ionizing radiation with more than 1 mSv in the previous 12 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline differences in synaptic density. | Data analysis will be done when all subjects have undergone the baseline evaluation.
  Baseline differences in (regional) synaptic density between premanifest HD and controls.
Baseline differences in brain volume. | Data analysis will be done when all subjects have undergone the baseline evaluation.
  Baseline differences in (regional) brain volume between premanifest HD and controls.
Differences in the rate of decline of synaptic density. | Data analysis will be done when all subjects have undergone the 2-year follow-up evaluation.
  * Differences in the rate of decline of (regional) synaptic density between patients and controls.
  * Sensitivity to change for synaptic density.
Differences in the rate of decline of volumetric MRI. | Data analysis will be done when all subjects have undergone the 2-year follow-up evaluation.
  * Differences in the rate of decline of (regional) brain volumes between patients and controls.
  * Sensitivity to change for (regional) brain volumes.

SECONDARY OUTCOMES:
Baseline correlations between clinical scores and regional synaptic density or brain volume. | Data analysis will be done when all subjects have undergone the baseline evaluation.
  Correlations between clinical scores and regional synaptic density or regional volume loss in the patient group at baseline.
Correlations between progression of the clinical scores and decline of synaptic density or brain volume. | Data analysis will be done when all subjects have undergone the 2-year follow-up evaluation.
  Correlations between progression of the clinical scores and decline of synaptic density or regional volume loss in the patient group, after longitudinal follow up of 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided